CLINICAL TRIAL: NCT00897702
Title: Molecular Mechanisms of Clinical Resistance to Targeted Therapy Among Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-163; MSKCC-06163
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; male breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Blood Specimen Collection; Immunoenzyme Techniques; Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue and blood

INTERVENTIONS:
Other: Blood draw — A single 10ml tube of blood will also be obtained for a comparison of patient's normal DNA for genomic analyses either at the time of the procedure or at a followup appointment if feasible.
Other: immunoenzyme technique
Procedure: biopsy
Procedure: histopathologic examination

SUMMARY:
The purpose of this study is to learn why certain drugs stop working in patients.In lab studies, tumors become resistant in several ways. Specific molecules seem to change and this may be why therapy stops working. However, we do not know if the same molecules change in patients. This study is being done to see if they do change. If we learn more about how patients become resistant, we may be able to offer better treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Diagnosed with breast cancer.
* Patient must be able to consent to a biopsy
* Patient must be able to safely undergo a secondary biopsy, if needed.

Cohort 1

* Patients who previously received treatment with anti-HER2 therapy (including trastuzumab, pertuzumab, TDM1, lapatinib, neratibin, or DS8201) as part of adjuvant chemotherapy and now have progressive or recurrent breast cancer or, patients who previously (or currently) received anti-HER2 therapy as part of a regimen for metastatic breast cancer and subsequently experienced.
* Evidence of disease progression or recurrence after prior therapy (e.g. radiologic progression by RECIST criteria or new metastasis).
* Prior tumor biopsy (may be original) defined as HER2+ by amplification by FISH (>1.9 gene copy number) or IHC 3+.

Cohort 2

* Patients who previously received treatment with hormonal therapy (including aromatase inhibitors or SERMs or SERDs) as a part of adjuvant therapy and now have progressive or recurrent breast cancer or patients who previously (or currently) receive hormonal therapy as part of a regimen for metastatic breast cancer and subsequently experienced evidence of disease progression.

Cohort 3

* Patients not eligible for Cohorts 1 or 2.

Exclusion Criteria:

* Patients who are unable to consent to a biopsy.
* Patients for whom a repeat biopsy would be medically unsafe

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2007-01-09 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
To look for mutations in druggable oncogenic pathways in tumors progressing on anti-HER2 therapy or hormonal therapy | 3 years
To characterize the activity of the PI3K signaling pathway in progressive breast tumors using proteomic methods | 3 years
To develop new laboratory models of treatment refractory breast cancer from human tumor specimens | 3 years

SECONDARY OUTCOMES:
To look for mutations in druggable oncogenic pathways in tumor progressing on breast cancer targeted therapies | 3 years
To evaluate dynamic proteomic changes in response to inhibition of the RTK/PI3K/ATK/mTOR pathway. | 3 years
To characterize the genetic heterogeneity of progressive, metastatic tumors using next generation sequencing | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sarat Chandarlapaty, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT00897702/ICF_000.pdf